CLINICAL TRIAL: NCT02693145
Title: Cooperative Re-Engagement Controlled Trial (CoRECT)
Acronym: CoRECT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centers for Disease Control and Prevention (U.S. Federal Agency)
Collaborators: Connecticut State, Department of Mental Health and Addiction Services (Other Government); Massachusetts Department of Health (Other Government); Philadelphia Department of Public Health (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: FOA PS14-001
Record Dates: First submitted 2016-02-23; First posted 2016-02-26 (Estimated); Last update posted 2021-02-21 (Actual); Status verified 2021-02

CONDITIONS: Human Immunodeficiency Virus
Keywords: HIV/AIDS; re-engagement in care; data to care
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- standard of care (SOC) arm (No Intervention): Individuals found to be out of HIV medical care will receive standard of care to re-engage. This will not include use of disease intervention specialist to locate and recruit back to HIV medical care or use of the Anti-Retroviral Treatment and Access to Services (ARTAS) intervention.
- Intervention arm (Experimental): Individuals randomized to the intervention arm will receive field services to locate, contact, and provide assistance to access HIV medical care. Intervention may include use of disease intervention specialist to locate and recruit back to HIV medical care or use of the Anti-Retroviral Treatment and Access to Services (ARTAS) intervention.
  Interventions: Other: Anti-Retroviral Treatment and Access to Services (ARTAS)

INTERVENTIONS:
Other: Anti-Retroviral Treatment and Access to Services (ARTAS) — Anti-Retroviral Treatment and Access to Services (ARTAS) is an individual-level, multi-session, time-limited intervention with the goal of linking recently diagnosed persons with HIV to medical care soon after receiving their positive test result. ARTAS is based on the Strengths-based Case Management (SBCM) model, which is rooted in Social Cognitive Theory (particularly self-efficacy) and Humanistic Psychology. SBCM is a model that encourages the client to identify and use personal strengths; create goals for himself/herself; and establish an effective, working relationship with the Linkage Coordinator (LC).
  Arms: Intervention arm

SUMMARY:
CoRECT will help identify the important components of a data-sharing partnership between health departments and HIV care providers, and determine the extent to which a health department intervention can increase the number of HIV-infected persons out-of-care who: (a) link to an HIV clinic; (b) remain in HIV medical care; (c) achieve HIV viral load suppression within 12 months; and (d) achieve durable HIV viral load suppression over 18 months. We will also measure the cost-effectiveness of this intervention in regards to improved health in the individuals (re)-engaged in HIV care and reductions in further HIV transmission in the community.

DETAILED DESCRIPTION:
Methods summary: Health departments will generate an out-of-care list using HIV laboratory surveillance data; collaborating clinics will concurrently generate out-of-care lists using appointment data. The combined out-of-care list will be reconciled by the health department and clinics, and discussed at monthly case conferences. All individuals determined to be out-of care will be randomized to receive either: (1) usual linkage and engagement in care services (standard of care [SOC]); or (2) an active health department field services intervention in addition to SOC. The active intervention activities will vary among jurisdictions; however all sites will include field services to locate, contact, and provide assistance, including a same-day appointment, to access HIV medical care.

Study design: Each site will enroll 600 out-of-care HIV-infected individuals (300 per arm) during a two-year enrollment period. An out-of-care individual will be defined as: (1) a person who has received HIV medical care at a CoRECT clinic and then disengages from care; or (2) a person with newly diagnosed HIV infection who has an appointment at a CoRECT clinic, but has not linked to medical care within 90 days.

Intervention: Individuals randomized to the intervention arm will receive field services to locate, contact, and provide assistance to access HIV medical care. Services provided as part of the intervention will vary by jurisdiction, but may include assistance with expedited medical appointments, transportation, access to community resources such as traditional case management, strengths-based case management, or financial incentives (Appendix A).

Primary outcomes: The following outcomes will be compared between out-of-care HIV-infected individuals receiving the study intervention to those receiving usual services:

1. Attend 1 clinic visit within 90 days;
2. Remain engaged in care, defined as 2 clinic visits at least 3 months apart within 12 months;
3. Achieve viral load suppression within 12 months;
4. Achieve durable viral load suppression, defined as 2 consecutive suppressed viral load results at least 3 months apart within 18 months

ELIGIBILITY:
Inclusion Criteria:

1. Residents within the health department jurisdiction who have received HIV medical care at a CoRECT clinic and then disengage by either of the following definitions:

   * Clinic definition: did not have a visit with a prescribing provider for 6 months.
   * Health department definition: no CD4 or viral load test result reported to health department surveillance for more than 6 months.
2. Residents within the health department jurisdiction with newly diagnosed HIV infection who have not linked to medical care within 90 days and have either:

   * Received, but did not attend, an appointment at a CoRECT clinic; or
   * Attended an enrollment visit but did not receive medical care at a CoRECT clinic.

Exclusion Criteria:

1. Deceased
2. Out of jurisdiction
3. Changed providers
4. Incarcerated

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1893 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2020-08 (Actual); Study Completion 2020-08 (Actual)

PRIMARY OUTCOMES:
Attend one clinic visit | within 90 days of randomization
  Patient will attend one clinical visit at CoRECT clinic to receive HIV medical care
Remain engaged in care | defined as 2 clinic visits at least 3 months apart within 12 months
  Two or more medical visits at least 3 months apart within 12 months to demonstrate patient remains engaged in HIV medical care
Viral load suppression | within 12 months
  Does the patient achieve viral load suppression within 12 months of randomization
Achieve durable viral load suppression | defined as 2 consecutive suppressed viral load results at least 3 months apart within 18 months
  Achieve durable viral load suppression, defined as 2 consecutive suppressed viral load results at least 3 months apart within 18 months

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Connecticut Department of Public Health, Hartford, Connecticut
  - Massachusetts Department of Public Health, Boston, Massachusetts
  - Philadelphia Department of Health, Philadelphia, Pennsylvania

REFERENCES:
- [Background] The White House Office of National AIDS Policy. National HIV/AIDS Strategy. Available at: http://www.whitehouse.gov/administration/eop/onap/nhas. Accessed: 30 January 2015.
- [Background] Bradley H, Hall HI, Wolitski RJ, Van Handel MM, Stone AE, LaFlam M, Skarbinski J, Higa DH, Prejean J, Frazier EL, Patel R, Huang P, An Q, Song R, Tang T, Valleroy LA. Vital Signs: HIV diagnosis, care, and treatment among persons living with HIV--United States, 2011. MMWR Morb Mortal Wkly Rep. 2014 Nov 28;63(47):1113-7. PMID 25426654
- [Background] Skarbinski J, Rosenberg E, Paz-Bailey G, Hall HI, Rose CE, Viall AH, Fagan JL, Lansky A, Mermin JH. Human immunodeficiency virus transmission at each step of the care continuum in the United States. JAMA Intern Med. 2015 Apr;175(4):588-96. doi: 10.1001/jamainternmed.2014.8180. PMID 25706928
- [Background] Gardner LI, Metsch LR, Anderson-Mahoney P, Loughlin AM, del Rio C, Strathdee S, Sansom SL, Siegal HA, Greenberg AE, Holmberg SD; Antiretroviral Treatment and Access Study Study Group. Efficacy of a brief case management intervention to link recently diagnosed HIV-infected persons to care. AIDS. 2005 Mar 4;19(4):423-31. doi: 10.1097/01.aids.0000161772.51900.eb. PMID 15750396
- [Background] Gardner LI, Marks G, Craw JA, Wilson TE, Drainoni ML, Moore RD, Mugavero MJ, Rodriguez AE, Bradley-Springer LA, Holman S, Keruly JC, Sullivan M, Skolnik PR, Malitz F, Metsch LR, Raper JL, Giordano TP; Retention in Care Study Group. A low-effort, clinic-wide intervention improves attendance for HIV primary care. Clin Infect Dis. 2012 Oct;55(8):1124-34. doi: 10.1093/cid/cis623. Epub 2012 Jul 24. PMID 22828593
- [Background] Gardner LI, Giordano TP, Marks G, Wilson TE, Craw JA, Drainoni ML, Keruly JC, Rodriguez AE, Malitz F, Moore RD, Bradley-Springer LA, Holman S, Rose CE, Girde S, Sullivan M, Metsch LR, Saag M, Mugavero MJ; Retention in Care Study Group. Enhanced personal contact with HIV patients improves retention in primary care: a randomized trial in 6 US HIV clinics. Clin Infect Dis. 2014 Sep 1;59(5):725-34. doi: 10.1093/cid/ciu357. Epub 2014 May 15. PMID 24837481
- [Background] Dombrowski JC. Testing, Linkage and Retention in Care: Getting Control of the Cascade in Seattle. National Summit on HIV and Viral Hepatitis Diagnosis, Prevention, and Access to Care, Washington, DC, November 26-8, 2012.
- [Background] Udeagu CC, Webster TR, Bocour A, Michel P, Shepard CW. Lost or just not following up: public health effort to re-engage HIV-infected persons lost to follow-up into HIV medical care. AIDS. 2013 Sep 10;27(14):2271-9. doi: 10.1097/QAD.0b013e328362fdde. PMID 23669157
- [Background] Cohen MS, Chen YQ, McCauley M, Gamble T, Hosseinipour MC, Kumarasamy N, Hakim JG, Kumwenda J, Grinsztejn B, Pilotto JH, Godbole SV, Mehendale S, Chariyalertsak S, Santos BR, Mayer KH, Hoffman IF, Eshleman SH, Piwowar-Manning E, Wang L, Makhema J, Mills LA, de Bruyn G, Sanne I, Eron J, Gallant J, Havlir D, Swindells S, Ribaudo H, Elharrar V, Burns D, Taha TE, Nielsen-Saines K, Celentano D, Essex M, Fleming TR; HPTN 052 Study Team. Prevention of HIV-1 infection with early antiretroviral therapy. N Engl J Med. 2011 Aug 11;365(6):493-505. doi: 10.1056/NEJMoa1105243. Epub 2011 Jul 18. PMID 21767103
- [Derived] Macharaviani E, Altice FL, Shrestha R, Truebig J, Carroll C, Nichols L, Ahmad B, Copenhaver M, Villanueva M. Disease Intervention Specialist Field Experience in Re-engaging Out-of-Care People with HIV in Project CoRECT: A Mixed Methods Study. AIDS Behav. 2025 Aug;29(8):2451-2460. doi: 10.1007/s10461-025-04707-w. Epub 2025 Apr 10. PMID 40205311
- [Derived] Machavariani E, Miceli J, Altice FL, Fanfair RN, Speers S, Nichols L, Jenkins H, Villanueva M. Using Data-To-Care Strategies to Optimize the HIV Care Continuum in Connecticut: Results From a Randomized Controlled Trial. J Acquir Immune Defic Syndr. 2024 May 1;96(1):40-50. doi: 10.1097/QAI.0000000000003391. PMID 38324241
- [Derived] Elder H, Lang SG, Villanueva M, John B, Roosevelt K, Altice FL, Brady KA, Gibson B, Buchelli M, DeMaria A, Randall LM. Using the exploration, preparation, implementation, sustainment (EPIS) framework to assess the cooperative re-engagement controlled trial (CoRECT). Front Public Health. 2023 Dec 1;11:1223149. doi: 10.3389/fpubh.2023.1223149. eCollection 2023. PMID 38106893
- [Derived] O'Shea J, Fanfair RN, Williams T, Khalil G, Brady KA, DeMaria A Jr, Villanueva M, Randall LM, Jenkins H, Altice FL, Camp N, Lucas C, Buchelli M, Samandari T, Weidle PJ. The Cooperative Re-Engagement Controlled Trial (CoRECT): Durable Viral Suppression Assessment. J Acquir Immune Defic Syndr. 2023 Jun 1;93(2):134-142. doi: 10.1097/QAI.0000000000003178. PMID 36812382